CLINICAL TRIAL: NCT03950778
Title: The Effect of Albumin Supplementation on the Inflammatory and Oxidative Stress Markers in Septic Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Upecs-UP-MS-ICU-Albumin
Record Dates: First submitted 2019-04-16; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Albumin Supplementation; Albumin Therapy; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Septic patients receiving albumin replacement (Active Comparator): Septic patients receiving albumin replacement 20 ml Inj Human Albumin 20% -3x100 ml- 3 day
  Interventions: Drug: Human albumin
- Septic patients not receiving albumin replacement (No Intervention)

INTERVENTIONS:
Drug: Human albumin — Patients are divided into 2 groups by envelope randomization. In the treated group, albumin supplementation occurs up to a target of 30 g / l at the end of the test period at a maximum dose of 3 x 100 ml, and no albumin is added above the control value of 20 g / l. Patients with albumin below 20 g / l in the control group are excluded from the study and albumin supplemented. Blood samples are taken directly at the intensive care class, and at the same time on the following days. Urine was collected for 24 hours. The kinetics of the parameters are examined for five days.
  Arms: Septic patients receiving albumin replacement

SUMMARY:
There is currently no uniform target for serum albumin levels in some pathological conditions, but recent studies have shown that serum albumin concentrations, disease severity, and mortality rates have been linked. Although the exact mechanism is unclear, serum albumin levels may have a protective effect on the potential antioxidant effect of maintaining physiological homeostasis and its anti-inflammatory effects. The indication and efficacy of parenteral albumin therapy in the care of patients in critical condition has long been a hot topic. Although previous mortality endpoint studies were negative, it is not certain that they can be used clearly in intensive care. According to earlier research, albumin is a very important circulating antioxidant. It is believed that early suplementattion of albumin may have a beneficial effect on oxidative stress and inflammation in septic patients.

The aim of our study is to investigate changes in parameters (inflammation, oxidative stress) that can be directly influenced by the administration of albumin in septic cases in need of intensive care. Also in our earlier, relatively small number of studies, chemiluminescence analysis of non-enzymatic total antioxidant capacity showed an increase in total antioxidant capacity in septic patients. The proposed study may also clarify the background of pathophysiological changes behind this phenomenon.

DETAILED DESCRIPTION:
There is currently no uniform target for serum albumin levels in some pathological conditions, but recent studies have shown that serum albumin concentrations, disease severity, and mortality rates have been linked. Although the exact mechanism is unclear, serum albumin levels may have a protective effect on the potential antioxidant effect of maintaining physiological homeostasis and its anti-inflammatory effects. The indication and efficacy of parenteral albumin therapy in the care of patients in critical condition has long been a hot topic. Although previous mortality endpoint studies were negative, it is not certain that they can be used clearly in intensive care. According to earlier research, albumin is a very important circulating antioxidant. It is believed that early suplementattion of albumin may have a beneficial effect on oxidative stress and inflammation in septic patients.

The aim of our study is to investigate changes in parameters (inflammation, oxidative stress) that can be directly influenced by the administration of albumin in septic cases in need of intensive care. Also in our earlier, relatively small number of studies, chemiluminescence analysis of non-enzymatic total antioxidant capacity showed an increase in total antioxidant capacity in septic patients. The proposed study may also clarify the background of pathophysiological changes behind this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Primarily, patients with sepsis or septic shock are enrolled into patients who are admitted to an intensive care class or who become septic in the intensive care unit (based on the sepsis definition).

Exclusion Criteria:

* Under 18 years old
* documented treatment or co-morbidity affecting the immune response: malignant hematological disease
* chronic steroid use,
* biological therapy,
* taking immunosuppressive drugs after organ transplantation,
* end stage tumor disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The effect of albumin supplementation on PCT level | 24 months
  The effect of albumin supplementation on the inflammatory and oxidative stress marker PCT will be assesed
The effect of albumin supplementation on CRP level | 24 months
  The effect of albumin supplementation on the inflammatory and oxidative stress marker CRP will be assesed
The effect of albumin supplementation on serum- total protein concentration | 24 months
  The effect of albumin supplementation on the inflammatory and oxidative stress markers total protein will be assesed
The effect of albumin supplementation on albumin concentration | 24 months
  The effect of albumin supplementation on the inflammatory and oxidative stress marker albumin will be assesed

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - University of Pécs Department of Anaesthesiology and Intensive Therapy, Pécs, Ifjúság Str 13.
  - Universitty of Pecs Department of Anaesthesiology and Intensive Therapy, Pécs, Ifjúság Str.13.

IPD SHARING:
Plan to Share IPD: Undecided